CLINICAL TRIAL: NCT03540771
Title: Introducing Palliative Care (PC) Within the Treatment of End Stage Liver Disease (ESLD): A Cluster Randomized Controlled Trial
Brief Title: Introducing Palliative Care (PC) Within the Treatment of End Stage Liver Disease (ESLD)
Acronym: PAL-LIVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Manisha Verma, Director, Research, Department of Medicine, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00092149
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: End Stage Liver Disease; Decompensated Cirrhosis of Liver
Keywords: palliative care; hepatology; decompensated cirrhosis
MeSH Terms: conditions — End Stage Liver Disease | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Model 1: Consultative Palliative Care (i.e. direct access to Palliative Care provider), versus Model 2: Trained Hepatologist- led PC intervention (i.e. a hepatologist will receive formal training to deliver Palliative Care services)
Masking Description: The study investigators were masked to comparative outcomes measures until the study was completed and database was locked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Model 1: Consultative Palliative Care (Active Comparator): Direct access to Palliative Care provider, who will offer palliative care to patients and caregivers, as guided by a standard PC (palliative care) checklist.
  Interventions: Other: Palliative Care
- Model 2: Trained Hepatologist- led PC (Active Comparator): A hepatologist will receive formal training to deliver Palliative Care (PC) services, and will offer palliative care to patients and caregivers following the same PC checklist as in Model 1
  Interventions: Other: Palliative Care

INTERVENTIONS:
Other: Palliative Care — The intervention will comprise an approach to render palliative care, as taught to hepatologists through an on-line learning platform, and as delivered by PC providers as routine care. The elements of the intervention, which will be guided by a checklist and implemented over the course of interactions with the patient and caregivers at the initial, 1, 2, and 3 month visits, to include:
  1. Patient/caregiver understanding of diagnosis, illness and prognosis
  2. Symptom assessment and management
  3. Psychosocial assessment and management
  4. Distress screening and management
  5. Discussion of goals of care
  6. Advanced directives

SUMMARY:
This is a comparative effectiveness study of two pragmatic models aiming to introduce palliative care for end stage liver disease patients. The 2 comparators are:

Model 1: Consultative Palliative Care (i.e. direct access to Palliative Care provider), Model 2: Trained Hepatologist- led PC intervention (i.e. a hepatologist will receive formal training to deliver Palliative Care services)

Primary Outcome: The change in quality of life from baseline to 3 months post enrollment as assessed by FACT-Hep (Functional Assessment of Cancer Therapy- Hepatobiliary).

Primary Hypothesis: Compared to consultative PC, the trained hepatologist-led PC for ESLD patients will show superior primary outcome. In the event of nonsignificant superiority, the trained hepatologist-led PC led will show non-inferiority (NI) by ruling out a 4-point reduction (NI margin) in mean of the primary outcome as compared to the consultative PC.

Power: The study has 83.2% power to detect minimal clinically important difference (MCID) of 9 points in mean of the primary outcome between the two randomized arms. We have 79.2% power for the noninferiority hypothesis, under assumption that the trained hepatologist-led PC arm performs better than the consultative PC arm by half of the above MCID.

Setting: 19 Clinical Centers across US are recruited to participate in this study.

Qualitative nested study will interview patients, caregivers and providers to assess their experiences with participating in the palliative care trial.

DETAILED DESCRIPTION:
This is a two armed comparative effectiveness cluster randomized controlled trial (RCT), to assess the effectiveness of two pragmatic PC models for patients with ESLD (Consultative PC vs. Trained hepatologist led PC). To prevent bias at the level of providers, randomization will take place at the level of clinical centers; however patients will be the unit of inference. There is no standard of care arm.

Embedded within this cluster-RCT is a qualitative study will be undertaken to evaluate the patient/caregiver experiences in the two PC models, using semi structured interviews.

To execute this project, we have identified 19 clinical centers to participate; 8 Veterans Health Administration (VHA) systems and 11 non-VHA, Academic Medical Centers.

Comparative Approaches:

1. Consultative PC led approach (Model 1): The PC model will include: 1) routine PC consults, using a standardized checklist , 2) in-person or telehealth visits at initial, 1, 2 and 3 months. .
2. Trained hepatologist led PC (Model 2): The Hepatologist Led PC model will comprise: 1) Hepatologist training (through E Learning modules), and 2) in person or telehealth visits utilizing the same PC checklist as utilized in Model 1. The study visits will occur at initial, 1, 2 and 3 months i.e. similar to Model 1 and follow the same visit specified agenda.

Study visits in both models could occur in-person or telehealth based, especially during in-person visit restrictions due to COVID pandemic.

Adult patients with end stage liver disease and their caregivers 18 years of age or older will be enrolled.

Primary Outcome: The change in quality of life from baseline to 3 months post enrollment as assessed by FACT-Hep (Functional Assessment of Cancer Therapy- Hepatobiliary).

Primary Hypothesis: Compared to consultative PC, the trained hepatologist-led PC for ESLD patients will show superior primary outcome. In the event of nonsignificant superiority, the trained hepatologist-led PC led will show non-inferiority (NI) by ruling out a 4-point reduction (NI margin) in mean of the primary outcome as compared to the consultative PC.

Power: The study has 83.2% power to detect clinically important difference (MCID) of 9 points in mean of the primary outcome between the two randomized arms. We have 79.2% power for the noninferiority hypothesis, under assumption that the trained hepatologist-led PC arm performs better than the consultative PC arm by half of the above MCID.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients were adults (≥18 years) with:

1. cirrhosis and a decompensation event indicative of ESLD (such as ascites, variceal bleeding or hepatic encephalopathy) within the prior 6 months, or
2. hepatocellular cancer (HCC) except Barcelona Stage D, or multifocal HCC (as defined by standard guidelines and confirmed by treating hepatologist).

Additional inclusion criteria included English literacy and the capacity to complete study assessments.

Exclusion criteria were hepatologist assessed life expectancy <6 months, prior liver transplantation, anticipated liver transplantation within 3 months, inability to consent, or receipt of PC within the previous three months.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1494 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Verma, MD, MPH, Principal Investigator — Albert Einstein Healthcare Network; Victor Navarro, MD, Principal Investigator — Albert Einstein Healthcare Network
Locations (19):
- United States (19):
  - University of Alabama, Birmingham, Alabama
  - Banner Health- University Medical Center, Phoenix, Arizona
  - UCSF Fresno, Fresno, California
  - Loma Linda Unversity Health, Loma Linda, California
  - VA West Haven, West Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Miami VA Medical Center, Miami, Florida
  - Indiana University, Indianapolis, Indiana
  - VA Boston, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Kansas City VA Medical Center, Kansas City, Missouri
  - VA New York Harbor, Brooklyn, New York
  - VA Bronx, The Bronx, New York
  - UNC Liver Center, Chapel Hill, North Carolina
  - Durham V.A. Medical Center, Durham, North Carolina
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verma M, Tapper EB, Singal AG, Navarro V. Nonhospice Palliative Care Within the Treatment of End-Stage Liver Disease. Hepatology. 2020 Jun;71(6):2149-2159. doi: 10.1002/hep.31226. PMID 32167615
- [Background] DeNofrio JC, Verma M, Kosinski AS, Navarro V, Taddei TH, Volk ML, Bakitas M, Ramchandran K. Palliative Care Always: Hepatology-Virtual Primary Palliative Care Training for Hepatologists. Hepatol Commun. 2022 Apr;6(4):920-930. doi: 10.1002/hep4.1849. Epub 2021 Oct 31. PMID 34719137
- [Background] Verma M, Bakitas MA. Creating Effective Models for Delivering Palliative Care in Advanced Liver Disease. Curr Hepatol Rep. 2021;20(2):43-52. doi: 10.1007/s11901-021-00562-0. Epub 2021 Apr 10. PMID 33868897
- [Derived] Hoppmann N, Bakitas M, Stockdill M, DeNofrio J, Navarro V, Verma M. Palliative Care for Advanced Liver Disease: Hepatology and Palliative Care Specialists Experiences. J Pain Symptom Manage. 2026 Jan;71(1):157-167. doi: 10.1016/j.jpainsymman.2025.09.028. Epub 2025 Oct 8. PMID 41072740
- [Derived] Verma M, Kosinski AS, Volk ML, Taddei T, Ramchandran K, Bakitas M, Green K, Green L, Navarro V. Introducing Palliative Care within the Treatment of End-Stage Liver Disease: The Study Protocol of a Cluster Randomized Controlled Trial. J Palliat Med. 2019 Sep;22(S1):34-43. doi: 10.1089/jpm.2019.0121. PMID 31486722
- See also: PCORI web release — https://www.pcori.org/research-results/2017/comparing-two-ways-offer-palliative-care-improve-quality-life-patients-end-stage-liver-disease

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients and caregivers separately. 935 Patients ( 516 in Model 1 and 419 in Model 2) and 559 caregivers (310 in Model 1 and 249 in Model 2) were enrolled. Recruitment occured from January 2019 to March 2025, with completion of data collection and database lock by June 30, 2025. Each row represents the patient and caregiver characteristics based on the actual enrollment numbers.
Pre-assignment Details: This study consented and enrolled patients and caregivers separately. 935 Patients ( 516 in Model 1 and 419 in Model 2) and 559 caregivers (310 in Model 1 and 249 in Model 2) were enrolled.
Units Other Than Participants: Clinical Centers
Groups:
- Model 1: Consultative Palliative Care: Direct access to Palliative Care provider, who will offer palliative care to patients and caregivers, as guided by a standard PC (palliative care) checklist.
  Palliative Care: The intervention will comprise an approach to render palliative care, as taught to hepatologists through an on-line learning platform, and as delivered by PC providers as routine care. The elements of the intervention, which will be guided by a checklist and implemented over the course of interactions with the patient and caregivers at the initial, 1, 2, and 3 month visits, to include:
  1. Patient/caregiver understanding of diagnosis, illness and prognosis
  2. Symptom assessment and management
  3. Psychosocial assessment and management
  4. Distress screening and management
  5. Discussion of goals of care
  6. Advanced directives
- Model 2: Trained Hepatologist- Led PC: A hepatologist will receive formal training to deliver Palliative Care (PC) services, and will offer palliative care to patients and caregivers following the same PC checklist as in Model 1
  Palliative Care: The intervention will comprise an approach to render palliative care, as taught to hepatologists through an on-line learning platform, and as delivered by PC providers as routine care. The elements of the intervention, which will be guided by a checklist and implemented over the course of interactions with the patient and caregivers at the initial, 1, 2, and 3 month visits, to include:
  1. Patient/caregiver understanding of diagnosis, illness and prognosis
  2. Symptom assessment and management
  3. Psychosocial assessment and management
  4. Distress screening and management
  5. Discussion of goals of care
  6. Advanced directives
Period: Overall Study
Arm/Group | Model 1: Consultative Palliative Care | Model 2: Trained Hepatologist- Led PC
Started | 826; 8 Clinical Centers (Eight Clinical Centers were assigned to Model 1 (Consultative PC). Number of Patients enrolled= 516; Number of Caregivers enrolled=310. Total number of participants= 826) | 668; 11 Clinical Centers (Eleven Clinical Centers were assigned to Model 2 (Trained Hepatologist led PC). Number of Patients enrolled= 419;Number of Caregivers enrolled in Model 2=249 Total number of participants= 668)
Completed | 558; 8 Clinical Centers (All centers completed the study for their enrolled participants. Number of Patients completed study intervention (3 months)=368; Number of Caregivers completed study intervention (3 months) =190 Total participants completed= 558) | 456; 11 Clinical Centers (All centers completed the study for their enrolled participants Number of Patients completed study intervention (3 months)=299; Number of Caregivers completed study intervention (3 months) =157 Total participants completed= 456)
Not Completed | 268; 0 Clinical Centers | 212; 0 Clinical Centers

BASELINE CHARACTERISTICS:
Population: The total study participants (1494) includes 935 patients (516 in Consultative PC and 419 in Trained Hepatologist led PC) and 559 caregivers (310 in Consultative PC and 249 in Trained Hepatologist led PC)
Groups:
- Total: Total of all reporting groups
Arm/Group | Model 1: Consultative Palliative Care | Model 2: Trained Hepatologist- Led PC | Total
Number analyzed (Participants) | 826 | 668 | 1494
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: This study enrolled patients and caregivers separately. Each row represents the patient and caregiver characteristics based on the actual enrollment numbers. Hence the number analyzed differes in each row and the overall represents- patients only (as patient outcomes are the primary outcomes for this trial)
  years
    Patients: number analyzed (Participants) | 516 | 419 | 935
    Patients | 64 (10) | 62 (10.4) | 63 (10.3)
    Caregivers: number analyzed (Participants) | 310 | 249 | 559
    Caregivers | 58 (14.2) | 58 (14.2) | 58 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This study enrolled patients and caregivers separately. Each row represents the patient and caregiver characteristics based on the actual enrollment numbers. Hence the number analyzed differes in each row and the overall represents- patients only (as patient outcomes are the primary outcomes for this trial)
  Participants
    Patients: number analyzed (Participants) | 516 | 419 | 935
    Patients: Female | 123 | 152 | 275
    Patients: Male | 393 | 267 | 660
    Caregivers (separate from patients): number analyzed (Participants) | 310 | 249 | 559
    Caregivers (separate from patients): Female | 244 | 186 | 430
    Caregivers (separate from patients): Male | 66 | 63 | 129
Race (NIH/OMB) [Count of Participants; unit: Participants] — We report the baseline measures for patients and caregivers separately. Population: Patients and caregiver race data are reported separately. Thank you.
  Participants
    Patient participants: number analyzed (Participants) | 516 | 419 | 935
    Patient participants: American Indian or Alaska Native | 7 | 4 | 11
    Patient participants: Asian | 7 | 4 | 11
    Patient participants: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Patient participants: Black or African American | 87 | 60 | 147
    Patient participants: White | 409 | 332 | 741
    Patient participants: More than one race | 0 | 0 | 0
    Patient participants: Unknown or Not Reported | 6 | 18 | 24
    Caregiver participants: number analyzed (Participants) | 310 | 249 | 559
    Caregiver participants: American Indian or Alaska Native | 2 | 2 | 4
    Caregiver participants: Asian | 7 | 3 | 10
    Caregiver participants: Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
    Caregiver participants: Black or African American | 50 | 30 | 80
    Caregiver participants: White | 248 | 198 | 446
    Caregiver participants: More than one race | 0 | 0 | 0
    Caregiver participants: Unknown or Not Reported | 0 | 16 | 16
FACT-Hep total score [Mean (Standard Deviation); unit: units on a scale] — FACT-Hep total score ranges from 0-180. Higher scores reflect better quality of life. Population: This questionnaire is completed by patient participants only. This is a disease specific quality of life instrument which applies to patients only.
  units on a scale
    number analyzed (Participants) | 516 | 419 | 935
    (all) | 118.2 (28.0) | 113.4 (28.1) | 116.1 (28.2)
Zarit Burden Interview- 12 [Mean (Standard Deviation); unit: units on a scale] — This is a short, validated instrument to measure caregiver burden. Higher scores reflect higher burden. Range 0-48. Population: This questionnaire is completed by caregiver participants only.
  units on a scale
    number analyzed (Participants) | 310 | 249 | 559
    (all) | 8.7 (8.2) | 10.0 (8.2) | 9.2 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life (QOL)
Description: FACT-Hep (Functional Assessment of Cancer Therapy- Hepatobiliary) will be used to assess QOL. This is a 45 item self-reported instrument. FACT-Hep total score is the primary outcome. The scores range from 0 to 180. Higher scores reflect better QOL.
  This measure is for patients only.
Time Frame: Mean change in FACT-Hep total score from baseline to 3 months
Population: Modified Intention to treatment population excludes patients who got a liver transplant or were transferred to Hospice within 3 months of enrollment (i.e. before completion of intervention).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Model 1: Consultative Palliative Care | Model 2: Trained Hepatologist- Led PC
Number analyzed (Participants) | 499 | 410
score on a scale | 7.02 [4.34 to 9.71] | 8.01 [5.38 to 10.65]

2. Secondary Outcome: Patient's Symptom Burden
Description: Modified Edmonton Symptom Assessment Scale (ESAS) evaluated 13 symptoms (tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, shortness of breath, muscle cramps, sexual function, sleep, itch, pain) on a 10-point scale, where 0 is no symptom and 10 is the maximum severity of symptom. The total score ranges from 0-130. Higher scores reflect higher symptom burden.
  This measure is for patients only.
Time Frame: Change in ESAS total score from baseline to 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Model 1: Consultative Palliative Care | Model 2: Trained Hepatologist- Led PC
Number analyzed (Participants) | 499 | 410
score on a scale | -5.31 [-7.59 to -3.02] | -7.52 [-9.89 to -5.15]

3. Secondary Outcome: Patient's Depression Severity
Description: PHQ-9 (Personal Health Questionnaire) is one of the very commonly used tools to assess severity of depression in different settings, and has 9 questions. Each question is rated on a 4 point scale, with total score ranging from 0 to 27. Higher scores reflects greater severity of depression. Scores from 0-4 equates to no depression, 5-9 mild, 10-14 moderate, 15-19 mod severe and >20 reflects severe depression.
  This measure is for patients only.
Time Frame: Change in PHQ-9 scores from baseline to 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Model 1: Consultative Palliative Care | Model 2: Trained Hepatologist- Led PC
Number analyzed (Participants) | 499 | 410
score on a scale | -0.90 [-1.49 to -0.31] | -1.18 [-1.78 to -0.57]

4. Secondary Outcome: Patient Satisfaction
Description: FAMCARE-P13 (Family Satisfaction with Cancer Care- Patient scale) is a brief validated instrument used to assess patient satisfaction with outpatient palliative care interventions. It consists of 13 questions, with Likert scale response options. Higher scores imply better satisfaction from the care received.
  This measure is for patients only.
Time Frame: Change in FAMCARE-P scores from baseline to 3 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Model 1: Consultative Palliative Care | Model 2: Trained Hepatologist- Led PC
Number analyzed (Participants) | 499 | 410
score on a scale | 0.91 [-0.15 to 1.96] | 3.37 [2.24 to 4.49]

5. Secondary Outcome: Distress
Description: Distress thermometer (DT) ranks level of distress from 0- 10, Higher scores reflect higher distress.
  This is for patients only.
Time Frame: Change in Distress from baseline to 3 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Model 1: Consultative Palliative Care | Model 2: Trained Hepatologist- Led PC
Number analyzed (Participants) | 499 | 410
score on a scale | -0.34 [-0.63 to -0.06] | -0.27 [-0.58 to 0.03]

6. Secondary Outcome: Goal Concordant Care Questionnaire/ GCC (Patients)
Description: There are two subscales which assess Goal Concordant Care (GCC):
  1. Goals of Care Conversations (GoC) (7 items scale), assessing the perceived extent to which providers have engaged the patient in the process of advance care planning (score range 0-10) and
  2. Care Concordant with Preferences (CCP) (4 items scale), measuring the perceived alignment of delivered care with patient preferences (score range 0-2).
  Higher values represent a better outcome. There is no total score for this measure, only subscale scores apply.
Time Frame: Change in GCC scales from baseline to 3 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Model 1: Consultative Palliative Care | Model 2: Trained Hepatologist- Led PC
Number analyzed (Participants) | 499 | 410
score on a scale
  Goals of Care Conversations (GoC) scale | 0.17 [0.08 to 0.26] | 0.35 [0.27 to 0.44]
  Care Concordant with Preferences (CCP) scale | 0.53 [0.35 to 0.70] | 0.71 [0.52 to 0.89]

7. Secondary Outcome: Caregiver Burden (Completed by the Caregivers of Patients Who Were Enrolled as a Dyad). Caregivers Were Consented Separately.
Description: Zarit Burden Interview-12 (ZBI-12) a short, validated instrument is extensively used for palliative care research in diverse populations. It has high internal consistency, reliability and convergent validity to assess caregiver burden. Higher score reflects higher caregiver burden. The score ranges from 0- 48.
  This measure is for caregivers only.
Time Frame: Change in ZBI-12 scores from baseline to 3 months
Population: Caregivers were enrolled separately. The study enrolled patients with caregivers or patients alone.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Model 1: Consultative Palliative Care | Model 2: Trained Hepatologist- Led PC
Number analyzed (Participants) | 296 | 240
score on a scale | -0.69 [-1.72 to 0.33] | 0.73 [-0.34 to 1.79]

8. Secondary Outcome: Caregiver Quality of Life
Description: PROMIS- 29 (Patient Reported Outcomes Measurement Information System) assess overall quality of life and is summarized as : Physical and Mental health summary scores. Range 0-100 for both. Higher scores reflect higher physical function but worse mental health (as higher scores reflect higher domain assessed).
  Here we report for caregivers only.
Time Frame: Change in caregiver QoL from baseline to 3 months
Population: Modified Intention to treatment population excludes caregivers whose patients who got a liver transplant or were transferred to Hospice within 3 months of enrollment (i.e. before completion of intervention).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Model 1: Consultative Palliative Care | Model 2: Trained Hepatologist- Led PC
Number analyzed (Participants) | 296 | 240
score on a scale
  Physical Health Summary Score | 0.19 [-0.43 to 0.82] | 0.18 [-0.47 to 0.84]
  Mental Health Summary Score | -0.10 [-1.14 to 0.94] | -0.49 [-1.59 to 0.62]

9. Secondary Outcome: Goal Concordant Care/ GCC (Caregivers)
Description: There are two subscales which assess Goal Concordant Care (GCC):
  1. Goals of Care Conversations (GoC) (7 items scale), assessing the perceived extent to which providers have engaged the patient in the process of advance care planning (score range 0-10) and
  2. Care Concordant with Preferences (CCP) (4 items scale), measuring the perceived alignment of delivered care with patient preferences (score range 0-2).
  Higher values represent a better outcome. There is no total score for this measure, only subscale scores apply.
  Here we report for caregivers.
Time Frame: Change in GCC from baseline to 3 months
Population: Modified Intention to treatment population excludes caregivers of patients who got a liver transplant or were transferred to Hospice within 3 months of enrollment (i.e. before completion of intervention).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Model 1: Consultative Palliative Care | Model 2: Trained Hepatologist- Led PC
Number analyzed (Participants) | 296 | 240
score on a scale
  Goals of Care Conversations (GoC) scale | 0.21 [0.09 to 0.32] | 0.45 [0.33 to 0.57]
  Care Concordant with Preferences (CCP) scale | 0.32 [0.06 to 0.58] | 0.87 [0.61 to 1.14]

10. Secondary Outcome: Mortality Over 12 Months.
Description: Number of Patients that Died from Baseline to 12 Month.
Time Frame: Survival over 12 months
Population: All enrolled patients are included in this analysis. We report the number of patients who died within 12 months from enrollment (as count of participants).
Measure: Count of Participants; unit: Participants
Arm/Group | Model 1: Consultative Palliative Care | Model 2: Trained Hepatologist- Led PC
Number analyzed (Participants) | 516 | 419
Participants | 84 | 81

ADVERSE EVENTS:
Time Frame: All patients were followed for 1 year from enrollment. All-Cause Mortality, Serious Adverse Events and Other Adverse Events data were monitored for patients only.
Description: There were no adverse events related to study intervention (i.e. receiving palliative care from palliative care specialists or hepatologists) reported for patients enrolled in the trial.
  Mortality data was collected for patients only. Mortality was unrelated to the study participation or study intervention in all cases.
Arm/Group | Model 1: Consultative Palliative Care | Model 2: Trained Hepatologist- Led PC
All-Cause Mortality (participants affected / at risk) | 84/516 | 81/419
Serious Adverse Events (participants affected / at risk) | 0/516 | 0/419
Other Adverse Events (participants affected / at risk) | 0/516 | 0/419

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol with detailed outcomes and procedures (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT03540771/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Detailed Statistical Analysis Plan (2025-04-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT03540771/SAP_001.pdf